CLINICAL TRIAL: NCT05953012
Title: A Multi-center, Open-Label, Phase 1, Single- and Multiple Ascending Dose Study to Assess Safety and Tolerability of PMC-403 in Subjects With Neovascular Age-related Macular Degeneration (nAMD).
Brief Title: Study to Assess Safety and Tolerability of PMC-403 in Subjects With Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmAbcine (Industry)
Collaborators: C&R Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMC403-A01
Record Dates: First submitted 2023-06-14; First posted 2023-07-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: PMC-403

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PART 1- SAD (Experimental): The SAD part of the study will be conducted in a step-wise manner for a total of 4 dose levels of PMC-403.
  * Dose level 1: 0.7 mg/eye, baseline(Day 0)
  * Dose level 2: 2 mg/eye, baseline(Day 0)
  * Dose level 3: 3 mg/eye, baseline(Day 0)
  * Dose level 4: 4 mg/eye, baseline(Day 0)
  Interventions: Drug: PMC-403
- PART 2- MAD (Experimental): Upon the end of the SAD part of the study, the MAD part is planned to be conducted in a step-wise manner for a total of 2 dose levels.
  * Dose level 1: 3 mg/eye, baseline(Day 0), Week 4(Day 28), Week 8(Day 56)
  * Dose level 2: 4 mg/eye, baseline(Day 0), Week 4(Day 28), Week 8(Day 56)
  Interventions: Drug: PMC-403

INTERVENTIONS:
Drug: PMC-403 — PMC-403 will be administered Intravitreal.
  Other Names: Monotherapy

SUMMARY:
This is a Phase 1 study, first-in-human (FIH), open label study to evaluate the safety, tolerability and identify the maximum tolerated dose (MTD) of PMC-403 and determine the recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
In this study, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) will be carried out in a sequential manner.

- PART 1- SAD

The SAD part of the study will be conducted in a step-wise manner for a total of 4 dose levels (0.7 mg, 2 mg, 3 mg, 4 mg). To each dose group, 3 subjects at minimum or 6 subjects at maximum will be recruited. In the SAD part, dose escalation will be performed up to 4 mg/eye (50 uL/eye) until the MTD is identified.

In the SAD part, a maximum of 24 participants are to be enrolled.

- PART 2- MAD

Upon the end of the SAD part of the study, the MAD part is planned to be conducted in a step-wise manner for a total of 2 dose levels (3 mg, 4 mg).

In the MAD part will begin with dose level 1 (3 mg). Subjects will be given a total of 3 doses of IP at 4-week intervals over a total period of 12 weeks and will be assessed for safety and tolerability according to study procedures. While a total of 6 subjects are to be recruited per dose group in the MAD part. Dose escalation will be performed up to 4 mg/eye (50 uL/eye) until the MTD is identified.

In the MAD part, a maximum of 12 participants are to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study participation, subjects must meet all of the following inclusion criteria.

* Criteria for the selection of the study eye

If both eyes meet the criteria, the study eye will be selected according to the following criteria:

1. The eye with lower (severer) best corrected visual acuity (BCVA) at baseline will be selected as the study eye.
2. If both eyes have the same BCVA, the right eye will be selected as the study.

   1. Male and female ≥50 years of age at the time of written informed consent.
   2. Treatment required, based on the judgment of the investigator, due to insufficient therapeutic efficacy despite ≥ 3 repeated doses of anti-vascular endothelial growth factor (anti-VEGF) intravitreal injection (IVT) for nAMD in the study eye, and the subject's agreement to receive the study drug instead of conventional standard therapy
   3. >12 weeks must have elapsed since the last dose of anti-VEGF IVT at the time of screening.
   4. Active subfoveal or parafoveal choroidal neovascularization (CNV)* confirmed by fundus fluorescein angiography (FFA), spectral domain-optical coherence tomography (SD-OCT), and IndoCyanine Green (ICG) angiography.

      *Active CNV (confirmed by the central reading center) is defined as the presence of subretinal fluid (SRF) or intraretinal fluid (IRF) in consequence of vascular leakage.
   5. The size of the entire lesion in the study eye (including blood, atrophy, fibrosis, and neovascularization) must be ≤ 9-disc areas, and the area of CNV in the study eye must account for ≥ 50% of the total area of the lesion, as confirmed by FFA and ICG angiography.
   6. BCVA measured in the study eye must be between ≥ 23 letters and ≤ 78 letters based on the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart (Snellen visual acuity 20/25 - 20/320).
   7. Voluntary written informed consent to study participation.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not eligible for study participation.

1. At the screening visit:

   1. Uncontrolled ocular hypertension (≥ 25 mmHg) despite drug therapy;
   2. Retinal pigment epithelium (RPE) tears involving the macula;
   3. Improvement in visual acuity is not expected due to scars, fibrosis, or atrophy involving the fovea;
   4. Presence of vitreous hemorrhage;
   5. Aphakia or absence of posterior capsule (with the exception of pseudophakic eyes treated with laser posterior capsulotomy);
   6. Presence of any causes of CNV other than nAMD, such as ocular histoplasmosis, trauma, pathological myopia, angioid streak, choroidal rupture, or uveitis; or
   7. Macular pathology that is unrelated to nAMD, but may affect visual acuity or study drug treatment (e.g., macular hole, epiretinal membrane, vitreomacular traction, macular telangiectasia, central serous chorioretinopathy, retinal vascular occlusion, etc.).
2. Any of the following conditions or medical history in either eye:

   1. Current or known history of at least moderate diabetic retinopathy or diabetic macular edema;
   2. Active intraocular or periocular infections or inflammations (e.g., infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, etc.); or
   3. History of idiopathic or autoimmune uveitis.
3. Any of the following systemic diseases:

   1. Unstable or serious cardiovascular disorders such as congestive heart failure (New York Heart Association Functional Class III or IV), ventricular tachycardia requiring continuous treatment, unstable angina pectoris, or critical limb ischemia;
   2. Uncontrolled hypertension with systolic or diastolic blood pressure > 160/100 mmHg;
   3. Stroke or myocardial infarction within 24 weeks prior to screening;
   4. Dementia or neurodegenerative disorders (e.g., Alzheimer's disease, Parkinson's disease) that might affect study results during the study period;
   5. History of malignant tumors within 5 years prior to screening; or
   6. Weakened immunity or requiring immunotherapy.
   7. Clinically significant liver/kidney disease or any of the following hematologic test results:

      * Serum creatinine ≥1.5 x upper limit of normal
      * Aspartate transaminase (AST) or alanine transaminase (ALT) ≥2 x upper limit of normal
4. Treatment with any of the following systemic drug therapy:

   1. Systemic anti-VEGF therapy within 12 weeks prior to baseline;
   2. Systemic corticosteroids for ≥2 consecutive weeks

      * ≤ 10 mg/day prednisolone or equivalent for less than 2 consecutive weeks will be allowed
      * Inhaled, nasal, and topical steroids will also be allowed
   3. Ongoing treatment with any drugs with potential toxicity to the lens, retina, and optic nerves (e.g., deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazines, vigabatrin, or ethambutol).
5. Any of the following medical history (surgical or procedural):

   1. Intraocular or periocular injection of corticosteroids (e.g., triamcinolone acetonide, etc.) to the study eye within 24 weeks prior to screening;
   2. Intraocular surgery or laser therapy (e.g., cataract surgery, laser posterior capsulotomy, etc.) to the study eye within 12 weeks prior to screening;
   3. Eyelid surgery within 4 weeks prior to screening;
   4. History of vitrectomy, glaucoma surgery, macular laser treatment, keratoplasty, or retinal detachment surgery; or
   5. History of treatment with radiotherapy around the study eye including radiation retinopathy
6. Any concurrent ophthalmic abnormalities that, based on the judgment of the investigator, may affect the assessment of safety and therapeutic efficacy or may need medical or surgical treatment during the study period (e.g., cloudy ocular media, optic neuropathy, amblyopia, etc.).
7. Hypersensitivity to any of the components of IP or to contrast agents used for FFA and ICG angiography.
8. Pregnant and/or breastfeeding women.
9. Men and women of childbearing potential who are unwilling to use adequate methods of contraception* or who are planning a pregnancy during the study period and for 12 weeks from the last dose of IP

   -Methods of contraception: hormone contraceptives (oral contraceptives, contraceptive patch, etc.), intrauterine device (IUD) (copper IUD, hormonal intrauterine system), double barrier method (both male [condom] and female [diaphragm, vaginal sponge, or cervical cap]), surgical sterilization (tubal sterilization, vasectomy, etc.)
10. Having participated in another clinical trial and treated with an IP within 12 weeks prior to screening
11. Distance vision test result of <0.1 for the fellow eye
12. Other reasons based on which individuals are determined by the investigator to be ineligible for study participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline upto 4 weeks
  To identify the maximum tolerated dose (MTD), and determine the recommended phase 2 dose (RP2D) of PMC-403 in patients with nAMD.
  MTD of PMC-403 will be calculated by incidence of DLT at 4 weeks from the first dosing of PMC-403.
Adverse events | Baseline upto 5 months
  For Treatment-emergent adverse events (TEAEs), Adverse Drug Reactions (ADRs), Serious Adverse Events (SAEs), Serious Adverse Drug Reactions (SADRs), and Adverse Events (AEs) leading to study withdrawal, number of subjects, incidence, number of events, and 95% two-sided confidence interval will be presented by dose group.
Vital Signs - Pulse Rate (beats/min) | Baseline upto 5 months
  At each visit, pulse rate will be measured. Vital signs collected will be assessed for change before and after IP dosing and/or change in normal/abnormal findings.
  By dose group, values at each time point will be presented with number of subjects, mean, standard deviation, median, minimum, and maximum; and change from baseline at each time point will be presented with number of subjects, mean, standard deviation, median, minimum, and maximum.
Vital Signs - body temperature | Baseline upto 5 months
  At each visit, body temperature will be measured. Vital signs collected will be assessed for change before and after IP dosing and/or change in normal/abnormal findings.
  By dose group, values at each time point will be presented with number of subjects, mean, standard deviation, median, minimum, and maximum; and change from baseline at each time point will be presented with number of subjects, mean, standard deviation, median, minimum, and maximum.
Vital Signs - systolic/diastolic blood pressure (mmHg) | Baseline upto 5 months
  At each visit, systolic/diastolic blood pressure will be measured. Vital signs collected will be assessed for change before and after IP dosing and/or change in normal/abnormal findings.
  By dose group, values at each time point will be presented with number of subjects, mean, standard deviation, median, minimum, and maximum; and change from baseline at each time point will be presented with number of subjects, mean, standard deviation, median, minimum, and maximum.
Laboratory tests - Hematology | Baseline upto 5 months
  Hematology will be performed at Visits 1, 2, 5, and 7 and at Follow-up Visits 8 and 9 in the SAD groups and at each visit in the MAD groups.
  The following Hematology parameters will be recorded: white blood cell (WBC), red blood cell (RBC), hemoglobin, hematocrit, platelet, WBC differential count (neutrophil, lymphocyte, monocyte, eosinophil, basophil)
  Test results collected will be assessed for change before and after IP dosing and/or change in normal/abnormal findings.
Laboratory tests - Blood chemistry | Baseline upto 5 months
  Blood chemistry will be performed at Visits 1, 2, 5, and 7 and at Follow-up Visits 8 and 9 in the SAD groups and at each visit in the MAD groups.
  The following Blood chemistry parameters will be recorded: glucose, aspartate transaminase (AST; SGOT), alanine transaminase (ALT; SGPT), total bilirubin, alkaline phosphatase (ALP), lactate dehydrogenase (LDH), total protein, albumin, blood urea nitrogen (BUN), creatinine, uric acid, sodium, potassium, chloride, calcium, phosphorus, C-reactive protein (CRP), HbA1c (to be tested at the screening visit only)
  Test results collected will be assessed for change before and after IP dosing and/or change in normal/abnormal findings.
Laboratory tests - Urinalysis | Baseline upto 5 months
  Urinalysis will be performed at Visits 1, 2, 5, and 7 and at Follow-up Visits 8 and 9 in the SAD groups and at each visit in the MAD groups.
  For continuous variables, values at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum; and change from baseline at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
  Additionally, test results collected will be assessed for change before and after IP dosing and/or change in normal/abnormal findings.
Laboratory tests - Blood coagulation | Baseline upto 5 months
  Blood coagulation will be performed at Visits 1, 2, 5, and 7 and at Follow-up Visits 8 and 9 in the SAD groups and at each visit in the MAD groups.
  For continuous variables, values at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum; and change from baseline at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
  Additionally, test results collected will be assessed for change before and after IP dosing and/or change in normal/abnormal findings.
Electrocardiogram (ECG) | Baseline upto 5 months
  Test results will be classified into normal/NCS and CS, and change from baseline at each time point and at the last visit will be presented with frequency and percentage in a shift table by dose group.
  The following ECG parameters will be recorded: heart rate, RR interval, HR interval, QTc interval and QRS interval.
Ophthalmologic examination - Slit lamp examination | Baseline upto 5 months
  Slit lamp examination measuring will be performed according to Schedule of Events.
  For continuous variables, values at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum. The ophthalmologic examination results will be assessed for change in normal/abnormal status before and after IP dosing.
Ophthalmologic examination - fundus examination | Baseline upto 5 months
  fundus examination measuring will be performed according to Schedule of Events. For continuous variables, values at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum. The ophthalmologic examination results will be assessed for change in normal/abnormal status before and after IP dosing.
Ophthalmologic examination - spectral domain-optical coherence tomography (SD-OCT) | Baseline upto 5 months
  SD-OCT will be performed according to Schedule of Events. For continuous variables, values at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum. The ophthalmologic examination results will be assessed for change in normal/abnormal status before and after IP dosing.
Ophthalmologic examination - intraocular pressure (IOP) | Baseline upto 5 months
  IOP will be performed according to Schedule of Events. During the study visits involving IP dosing (SAD: Visits 2, MAD: Visits 2, 5, 7), IOP will be measured a total of 3 times (once before dosing and twice after dosing).
  For continuous variables, values at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum. The ophthalmologic examination results will be assessed for change in normal/abnormal status before and after IP dosing.

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) | Baseline upto 5 months
  It is measured by early treatment of diabetic retinopathy study (ETDRS) chart at each point of visit.
  For BCVA will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum; and change from baseline at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
Change in central retinal thickness (CRT) | Baseline upto 5 months
  It is measured by SD-OCT at each point of visit.
  For CRT will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum; and change from baseline at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
Presence of intraretinal fluid (IRF) | Baseline upto 5 months
  It is measured by SD-OCT at each point of visit.
  For presence of IRF frequency, percentage, and 95% confidence interval will be presented by dose group.
Presence of subretinal fluid (SRF) | Baseline upto 5 months
  It is measured by SD-OCT at each point of visit.
  For presence of SRF frequency, percentage, and 95% confidence interval will be presented by dose group.
Presence of sub-RPE fluid | Baseline upto 5 months
  It is measured by SD-OCT at each point of visit.
  For presence of sub-RPE fluid frequency, percentage, and 95% confidence interval will be presented by dose group.
Change from baseline in choroidal neovascularization (CNV) lesion size as measured by Fundus Fluorescein Angiography (FFA) | Baseline upto 5 months
  FFA will be performed to measure the size of CNV lesions and to assess vascular leakage.
  For CNV lesion size will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum; and change from baseline at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
Change from baseline in CNV lesion size as measured by ICG angiography | Baseline upto 5 months
  ICG angiography will be performed to measure the size of CNV lesions and to assess vascular leakage.
  For CNV lesion size will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum; and change from baseline at each time point will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.

OTHER OUTCOMES:
Pharmacokinetic parameters - Area under the blood concentration-time curve (AUC) | Baseline upto 5 months
  Area under the blood concentration-time curve from baseline to each by time point.
  For PK endpoints, continuous variables will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
Pharmacokinetic parameters - Maximum blood concentration (Cmax) | Baseline upto 5 months
  Maximum concentration of drug by dose level.
  For PK endpoints, continuous variables will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
Pharmacokinetic parameters - Minimum blood concentration (Cmin) | Baseline upto 5 months
  Minimum concentration of drug by dose level.
  For PK endpoints, continuous variables will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
Pharmacokinetic parameters - Clearance (CL) | Baseline upto 5 months
  Clearance by dose level.
  For PK endpoints, continuous variables will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
Pharmacokinetic parameters - Volume of distribution (Vd) | Baseline upto 5 months
  Volume of distribution by dose level.
  For PK endpoints, continuous variables will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
Pharmacokinetic parameters - Half-life (T1/2) | Baseline upto 5 months
  Half-life by dose level.
  For PK endpoints, continuous variables will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum.
Immunogenicity parameters - ADA formation rate | Baseline upto 5 months
  Presence anti-drug antibody (ADA).
  For immunogenicity assessment, categorical variables will be presented by dose group with frequency, percentage, and 95% confidence interval.
Exploratory assessment -Change from baseline in CNV activity as measured by OCTA. | Baseline upto 5 months
  For OCTA assessment, continuous variables will be presented by dose group with number of subjects, mean, standard deviation, median, minimum, and maximum; and categorical variables will be presented by dose group with frequency, percentage, and 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: SeJoon Woo, Principal Investigator — Seoul National University Bundang Hospital
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Seoul, Bundang-gu
  - Yeungnam University, Daegu, Nam-gu
  - Yonsei University Health System, Seoul, Seodaemun-gu
  - ASAN Medical Center, Seoul, Songpa-gu

IPD SHARING:
Plan to Share IPD: No